CLINICAL TRIAL: NCT00657969
Title: Looking For Genetic and Environmental Risk Factors and Therapeutic Aspects in Cervical Artery Dissections
Acronym: CADISP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cervical Artery Dissections and Ischemic Stroke Patients - Consortium (Network)
Responsible Party: Dr. S Debette, Dr. C Grond-Ginsbach, Pr. D Leys, University Hospitals of Heidelberg and Lille
Other Study IDs: CADISP
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Cervical Artery Dissection; Stroke; Brain Infarction
Keywords: Polymorphism, genetic; Risk factors; Carotid Artery, Internal, Dissection; Vertebral Artery Dissection; Genetic predisposition; Outcome; Therapy
MeSH Terms: conditions — Stroke; Brain Infarction; Carotid Artery, Internal, Dissection; Vertebral Artery Dissection; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — DNA, plasma, serum

GROUPS / COHORTS (3):
- 1: CAD-group (Cervical Artery Dissection - group): consecutive patients with cervical artery dissection, with or without associated cerebral ischemia, hospitalized in one of the participating neurological centers; standardized inclusion and exclusion criteria apply
- 2: IS-group (Ischemic Stroke - Group): patients selected among consecutive patients hospitalized for an ischemic stroke without CAD, in the same centers as patients from group1, frequency-matched on age and gender with group1; standardized inclusion and exclusion criteria apply
- 3: HC-group (Healthy Control - Group): DNA of healthy individuals from existing DNA-databases will be used as controls for the Belgian, French, German and Swiss centers; the other centers are recruiting their own age- and sex-matched healthy controls; individuals from the 3 groups (CAD, IS and HC) are strictly matched on geographical origin in order to avoid stratification bias

SUMMARY:
The main purpose of this study is to look for genetic and environmental risk factors of cervical artery dissections, a major cause of ischemic stroke in young adults, in a large multicenter case-control trial

DETAILED DESCRIPTION:
Background: Cervical artery dissections (CAD) are a major cause of ischemic stroke, longstanding disability, and occasionally death in young adults. Several lines of evidence suggest genetic predisposition for CAD. Previous genetic studies were, however, inconclusive mainly due to insufficient numbers of patients. Our hypothesis is that CAD is a multifactorial disease caused by yet largely unidentified genetic variants and environmental factors, which may interact.

Aim: Our main aim is to look for genetic and environmental risk factors and gene-environment interactions potentially underlying CAD. In addition, therapeutic aspects are addressed in the setting of a multicenter registry.

Methods: We organized a multinational European network, CADISP (Cervical Artery Dissection and Ischemic Stroke Patients) which targets at increasing our knowledge on the pathophysiological mechanisms of this disease in a large, representative patient population. Within this network, we are aiming to perform a de novo genetic association analysis using both a genome-wide and a candidate gene approach. For this purpose, 1130 patients with CAD, 1130 patients with non-CAD ischemic stroke, and 1890 healthy controls are being recruited, and detailed clinical, laboratory, diagnostic, therapeutic and outcome data are being collected from all participating patients. We are expecting to reach the above numbers of subjects by the end of 2008. Analyses of the CADISP database might clarify a number of debated issues, including risk factors, stroke preventive treatment, and outcome predictors of CAD.

We present the strategy of a collaborative project searching for genetic risk factors of cervical artery dissections. We hope that the CADISP network will provide detailed and novel data on risk factors and treatment aspects of CAD.

ELIGIBILITY:
GROUP1:

Inclusion Criteria:

* Typical radiological aspect of dissection* in a cervical artery (carotid and/or vertebral);* Mural hematoma, pseudoaneurysm, long tapering stenosis, intimal flap, double lumen, or occlusion > 2 cm above the carotid bifurcation revealing a pseudo aneurysm or a long tapering stenosis after recanalisation
* Written informed consent

Exclusion Criteria:

* Purely intracranial dissection
* Dissection occurring after an endovascular procedure
* Known mendelian genetic disorder that can explain the dissection (e.g. vascular Ehlers-Danlos syndrome)

GROUP2:

Inclusion Criteria:

* Recent ischemic stroke
* No signs of CAD on extracranial duplex sonography and angiography (digital subtraction or magnetic resonance or CT), performed < 7 days after the stroke
* Written informed consent

Exclusion Criteria:

* Possible cerebral ischemia but normal cerebral imaging
* CAD cannot be ruled out (e.g.persistent arterial occlusion without mural hematoma)
* Endovascular or surgical procedure on the coronary, cervical or cerebral arteries during the 48 hours preceding the cerebral infarction
* Cardiopathies with a very high embolic risk (Mechanical prosthetic valves, mitral stenosis with atrial fibrillation, intracardiac tumor, infectious endocarditis, myocardial infarction<4 months)
* Arterial vasospasm following a subarachnoid haemorrhage
* Auto-immune disease possibly responsible for the cerebral infarction
* Known monogenic disease responsible for the cerebral infarction

GROUP3:

Inclusion criteria:

* Individuals from the general population without history of stroke, dissections in any artery, transient ischemic attack, coronary artery disease, peripheral artery disease
* Written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: groups 1 and 2: hospital-based, neurology departments group 3: community samples
Sampling Method: Non-Probability Sample
Enrollment: 4169 (Actual)
Dates: Start 2005-07; Primary Completion 2009-01 (Actual); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
association of genetic polymorphisms with cervical artery dissections | 2009

SECONDARY OUTCOMES:
association of environmental risk factors with cervical artery dissections | 2009
gene-environment interactions | 2009

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Debette, MD, PhD, Study Director — Department of Neurology (EA2691), University Hospital of Lille; Inserm, U744, Pasteur Institute, Lille, France; Caspar Grond-Ginsbach, PhD, Study Chair — Department of Neurology, University Hospital of Heidelberg, Germany; Didier Leys, MD PhD, Principal Investigator — Department of Neurology (EA2691), University Hospital of Lille, France
Locations (24):
- Sanatorio Allende, Córdoba, Argentina
- Belgium (2):
  - Department of Neurology, University Hospital of Brussels (ULB), Brussels
  - Department of Neurology, University Hospital of Leuven, Leuven
- Department of Neurology, Helsinki University Central Hospital, Helsinki, Finland
- France (7):
  - Department of Neurology, University Hospital of Amiens, Amiens
  - Department of Neurology, University Hospital of Besançon, Besançon
  - Department of Neurology, University Hospital of Dijon, Dijon
  - Department of Neurology, University Hospital of Lille, Lille
  - Inserm U744 Institut Pasteur de Lille, Lille
  - Department of Neurology, University Hospital Pitié-Salpêtrière, Paris
  - Department of Neurology, University Hospital Sainte-Anne, Paris
- Germany (4):
  - Rehabilitation Center, Schmieder-Klinik, Heidelberg
  - Department of Neurology, University Hospital of Heidelberg, Heidelberg
  - Department of Neurology, Hospital of Ludwigshafen, Ludwigshafen
  - Department of Neurology, University Hospital of Munich, Munich
- Italy (6):
  - Department of Neurology, University Hospital of Brescia, Brescia
  - Department of Neurology, Ospedale Maggiore Policlinico di Milano, Milan
  - Ospedale Milano San Raffaele, Milan
  - Department of Neurology, University Hospital Milano-Bicocca, Monza
  - Department of Neurology, University Hospital of Perugia, Perugia
  - Rehabilitation Center, IRCCS Santa Lucia, Roma, Rome
- Department of Neurology, University Hospital of Basel, Basel, Switzerland
- Department of Neurology, Cerrahpasa Medical Faculty, Istanbul University, Istanbul, Turkey (Türkiye)
- Department of Neuroscience, St George's University Hospital of London, London, United Kingdom

REFERENCES:
- [Background] Engelter ST, Brandt T, Debette S, Caso V, Lichy C, Pezzini A, Abboud S, Bersano A, Dittrich R, Grond-Ginsbach C, Hausser I, Kloss M, Grau AJ, Tatlisumak T, Leys D, Lyrer PA; Cervical Artery Dissection in Ischemic Stroke Patients (CADISP) Study Group. Antiplatelets versus anticoagulation in cervical artery dissection. Stroke. 2007 Sep;38(9):2605-11. doi: 10.1161/STROKEAHA.107.489666. Epub 2007 Jul 26. PMID 17656656
- [Background] Debette S, Metso TM, Pezzini A, Engelter ST, Leys D, Lyrer P, Metso AJ, Brandt T, Kloss M, Lichy C, Hausser I, Touze E, Markus HS, Abboud S, Caso V, Bersano A, Grau A, Altintas A, Amouyel P, Tatlisumak T, Dallongeville J, Grond-Ginsbach C; CADISP-group. CADISP-genetics: an International project searching for genetic risk factors of cervical artery dissections. Int J Stroke. 2009 Jun;4(3):224-30. doi: 10.1111/j.1747-4949.2009.00281.x. PMID 19659826